CLINICAL TRIAL: NCT03110068
Title: Nomogram for Preoperative Estimation of Microvascular Invasion Risk in Hepatocellular Carcinoma
Brief Title: Preoperative Estimation of Microvascular Invasion in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ming Kuang (Other)
Responsible Party: Sponsor-Investigator, Ming Kuang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: SYSU01-US-201701
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: microvascular invasion; serum biomarker; radiological feature; pathological differentiation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preoperative clinical/imaging features: In this project, there is only one study group which comprises of patients with Hepatocellular Carcinoma (HCC) who will undergo contrast-enhanced computed tomography (CECT) and contrast-enhanced ultrasound (CEUS).
  Interventions: Diagnostic Test: contrast-enhanced ultrasound; Diagnostic Test: contrast-enhanced computed tomography

INTERVENTIONS:
Diagnostic Test: contrast-enhanced ultrasound — The Aplio SSA-770A or Aplio 500 (Toshiba Medical Systems, Tokyo, Japan) equipped with a 375BT convex transducer (frequency range, 1.9 to 6.0 MHz). CHI is used with a mechanical index that ranged from 0.06 to 0.10. After activating CHI mode, a bolus injection of 2.4 ml of SonoVue (Bracco, Milan, Italy) is administered intravenously via an antecubital vein, followed immediately by a flush of 5 ml of normal saline solution. The targeted lesion should be observed continuously for 5 minutes, and the entire arterial and portal venous phases and several repetitions of the late phase are stored on the hard disk. The arterial, portal venous and late phases are defined as 0-30 s, 31-120 s and 121-360 s after the injection, respectively.
Diagnostic Test: contrast-enhanced computed tomography — The Aquilion 64-slice helical CT machine (Tokyo, Japan) is used. The imaging protocol for CT examinations is as follows: 0.5 mm × 64 mm collimation, 120 kV, 150-200 mAs for 64-slice helical CT examination. The standard triphasic scan procedure is used. An unenhanced helical sequence scan through the liver will be performed first; thereafter nonionic iodinated contrast material (Ultravist, Schering, Berlin, Germany) (1.5 mL/kg) will be administered via antecubital vein with power injection at a rate of 4 mL/s for 64-slice helical CT. The arterial phase sequence is obtained 25-32 s after contrast material administration, followed by a portal venous phase sequence 70 s after contrast agent administration.

SUMMARY:
Presence of microvascular invasion can be estimated preoperatively, by some clinical imaging features such as patient characteristics, serum biomarkers and radiological features. Contrast-enhanced ultrasonography (CEUS) and contrast-enhanced computed tomography (CECT) are routine preoperative conventional examinations for hepatocellular carcinoma (HCC) patients in China. Combining features of CEUS, CECT and clinical factors may improve preoperative MVI assessment. The purpose of this study is to construct a nomogram for preoperative MVI risk estimation with these possible factors.

ELIGIBILITY:
Inclusion Criteria:

* Asian patients aged 18～80 years old;
* With no preoperative anti-cancer treatment;
* Scheduled for radical liver resection;
* With both CEUS and CECT performed in 4 weeks before surgery;
* Postoperative histologically confirmed HCC;
* With sufficient surgical specimen for MVI detection (surgical margin ≥1cm);

Exclusion Criteria:

* Recurrent HCC or combined hepatocellular-cholangiocarcinoma;
* With extra-hepatic metastasis or macrovascular invasion;
* With incomplete clinical and imaging data;
* Non-radical resection;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between April 2017 and April 2019，all consecutive patients who will undergo curative resection (R0 resection) at the First Affiliated Hospital of Sun Yat-Sen University in Guangzhou, China, for HCC based on the modified WHO classification of tumors of the digestive system, are considered for inclusion. By the eligibility criteria stated below, MVI presentative rate is 30-42% in chinese HCC population as reported, and an estimated 400 patients will be needed for this study.
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2017-04-10 (Estimated); Primary Completion 2019-04-10 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Presence of microvascular invasion | Through patient enrollment completion, an average of 2 years
  Postoperative histologically confirmed microvascular invasion

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Director — Department of Medical Ultrasonics, Institute of Diagnostic and Interventional Ultrasound, The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, China.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lei Z, Li J, Wu D, Xia Y, Wang Q, Si A, Wang K, Wan X, Lau WY, Wu M, Shen F. Nomogram for Preoperative Estimation of Microvascular Invasion Risk in Hepatitis B Virus-Related Hepatocellular Carcinoma Within the Milan Criteria. JAMA Surg. 2016 Apr;151(4):356-63. doi: 10.1001/jamasurg.2015.4257. PMID 26579636
- [Background] Zhao H, Hua Y, Dai T, He J, Tang M, Fu X, Mao L, Jin H, Qiu Y. Development and validation of a novel predictive scoring model for microvascular invasion in patients with hepatocellular carcinoma. Eur J Radiol. 2017 Mar;88:32-40. doi: 10.1016/j.ejrad.2016.12.030. Epub 2016 Dec 27. PMID 28189206
- [Background] Feng LH, Dong H, Lau WY, Yu H, Zhu YY, Zhao Y, Lin YX, Chen J, Wu MC, Cong WM. Novel microvascular invasion-based prognostic nomograms to predict survival outcomes in patients after R0 resection for hepatocellular carcinoma. J Cancer Res Clin Oncol. 2017 Feb;143(2):293-303. doi: 10.1007/s00432-016-2286-1. Epub 2016 Oct 14. PMID 27743138